CLINICAL TRIAL: NCT01569360
Title: Randomised Open Study of the Efficiency and Tolerance of the Use of a Corset on the Respiratory Function of Spinal Cord Injury Patients
Brief Title: Study of the Impact of the Use of a Corset on the Respiratory Function of Patients With Spinal Cord Injury
Acronym: Garchoise
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P091121
Record Dates: First submitted 2012-03-26; First posted 2012-04-03 (Estimated); Last update posted 2013-12-19 (Estimated); Status verified 2012-02

CONDITIONS: Spinal Cord Injury; Tetraplegia; Paraplegia
Keywords: Spinal cord injury; Tetraplegia; Paraplegia; Respiratory function; Corset
MeSH Terms: conditions — Spinal Cord Injuries; Quadriplegia; Paraplegia; Respiratory Aspiration

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Corset (Active Comparator): the patients are assigned the use of a custome made corset during daytime
  Interventions: Device: Corset
- No corset (No Intervention): the patients do not use a corset during daytime

INTERVENTIONS:
Device: Corset — the patients are assigned the use of a custome made corset during daytime
  Arms: Corset

SUMMARY:
Corsets are often used in the management of patients with a spinal cord injury. They may help to rigidify the patients' trunk which might help some patients to sit upright; their use may also reduce the sensation of dyspnea some patients have while sitting upright. Due to spinal cord injury, abdominal muscles are weakened which can contribute to alter the respiratory function of the patients. But the corset by rigidifying the abdominal wall can improve the efficiency of the respiratory muscles in some patients and reduce dyspnea in the sitting position for some patients. However, when patients with spinal cord injury are followed over time, one can observe that some patients discontinue corset use. The investigators observed that the patients who pursue the corset use still have a significant improvement of their respiratory function with the corset while the patients who have discontinued the use have improved their respiratory function in the upright position (without the corset). As of now, the investigators do not know whether the use of the corset is discontinued because of a spontaneous improvement of the respiratory function or whether discontinuing the use of the corset may help to develop abdominal spasticity and therefore to improve respiratory function. The investigators seek to investigate this issue in order to optimize the management of patients who present spinal cord injury.

DETAILED DESCRIPTION:
Corsets are widely used in the management of spinal cord injury (SCI) patients. Their use provides a certain amount of rigidity to the trunk which may help some patients to maintain posture; they also may contribute when used in combination with contention to reduce orthostatic hypotension. Last, they may reduce dyspnea and improve respiratory tolerance while sitting. Indeed, patients with recent SCI worsen their respiratory function in the sitting position secondary to the hypotonia of abdominal muscles which places the diaphragm in a lower and less efficient position. The use of a corset rigidifies the abdominal wall and therefore improves the diaphragm contraction's efficiency leading to an improvement of vital capacity (VC) and a reduction of dyspnea in the sitting position. But although some patients continue to use a corset overtime, others discontinue its use. We recently observed that corset users presented an improvement of VC with corset use proportional to the improvement of VC observed in the supine position while patients who had discontinued its use did not exhibit a reduction of VC between the supine and the upright position suggesting that they presented a more rigid abdominal wall.

It is not known whether corset use discontinuation results from the spontaneous improvement respiratory function in the upright position or leads to the appearance of abdominal spasticity and to the improvement of respiratory function.

Therefore, we aim to study the effect of the long term corset use on SCI patients' respiratory function.

We will conduct a monocentric prospective open study of 56 SCI patients (SCI level ranging from C5 to T8 ASIA A or B) with a recent lesion (<4 months). The evolution of respiratory function and dyspnea with and without corset use will be studied over a 2 years period. An evaluation of spasticity overtime will also be conducted. After randomization (corset use or not) evaluation will be conducted after 3 months, 6 months, 1 year and 2 years and will include: pulmonary function test with and without corset in the upright position and in the supine position, blood gases, dyspnea scores in the different positions and spasticity assessment.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients ≥ 18ans
* Spinal cord injury with an ASIA score of A or B
* Spinal cord injury with an injury level from C5 to T8 (included)
* Initial injury < 4 months
* Previous medical examination
* Signed consent form

Exclusion Criteria:

* Unstable respiratory state (far from secondary infection or congestion episode)
* Refusal to participate to the study
* Pregnant or nursing women
* Previous corset use
* No affiliation to social security system
* Impossibility to sustain the sitting position for several weeks or months (due to skin sore or planned surgery …)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2012-03; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
Vital capacity in the upright and supine position | 1 hour
  Measurement of the vital capacity in the upright and supine position at day 0, 3 months, 6 months, 1 year and 2 years.

SECONDARY OUTCOMES:
Maximal respiratory pressures | 30 minutes
  Measurement of non invasive maximal respiratory inspiratory (Pimax) and expiratory (Pemax) pressures in the upright position at day 0, 3 months, 6 months, 1 year and 2 years.
Blood gases | 15 minutes
  Measurement of blood gases (PO2, PCO2 and O2 saturation) at rest at day 0, 3 months, 6 months, 1 year and 2 years.
Borg dyspnéa scale | 5 minutes
  evaluation of dyspnea in the supine and in the upright position with the Borg dyspnea scale at day 0, 3 months, 6 months, 1 year and 2 years.
Ashworth scale | 5 minutes
  Evaluation of spasticity with the Ashworth scale at day 0, 3 months, 6 months, 1 year and 2 years.
Penn scale | 5 minutes
  Evaluation of spasticity with the Penn scale at day 0, 3 months, 6 months, 1 year and 2 years.
Blood pressure | 5 minutes
  Evaluation blood pressure in the upright and in the supine position at day 0, 3 months, 6 months, 1 year and 2 years.

CONTACTS AND LOCATIONS:
Overall Officials: Helene Prigent, MD, PHD, Principal Investigator — Raymond Poincaré Hospital, Garches 92380 France